CLINICAL TRIAL: NCT02662205
Title: A Controlled Trial of Group Yoga Therapy at a College Counseling Center
Brief Title: Group Yoga Therapy at a College Counseling Center
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: We did not get adequate referrals.
Sponsor: Jenilee Sneed (Other)
Responsible Party: Sponsor-Investigator, Jenilee Sneed, Graduate Student, Oklahoma State University
Organization: Oklahoma State University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OKState
Record Dates: First submitted 2016-01-12; First posted 2016-01-25 (Estimated); Last update posted 2016-03-30 (Estimated); Status verified 2016-03

CONDITIONS: Psychological Distress; Mindfulness
MeSH Terms: interventions — Psychotherapy, Group

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Traditional Group (Active Comparator): Traditional process psychotherapy group
  Interventions: Other: Psychotherapy Group
- Yoga Therapy Group (Experimental): Psychotherapy group integrating yoga and process dialogue
  Interventions: Other: Yoga Therapy Group
- Yoga Class (Active Comparator): Yin yoga class
  Interventions: Other: Yoga class

INTERVENTIONS:
Other: Psychotherapy Group — Traditional process group
  Arms: Traditional Group
Other: Yoga class — Yin yoga class
  Arms: Yoga Class
Other: Yoga Therapy Group — Yoga psychotherapy group integrating yoga and process dialogue
  Arms: Yoga Therapy Group

SUMMARY:
Clients of the student counseling center at Oklahoma State University who are interested in participating in the study will be randomly assigned to a traditional process group, a yoga class, and a yoga therapy group. Outcome of the three conditions will be compared.

DETAILED DESCRIPTION:
Clients will be screened for appropriateness for group treatment and yoga. They will be randomly assigned to a traditional process group, a yoga class, and a yoga therapy group. Each condition will run concurrently for 8 weeks. Outcome measures will be administered before trial commencement and after the trial ends.

ELIGIBILITY:
Inclusion Criteria:

* Students at Oklahoma State University
* Appropriate for group therapy
* Physically capable of doing yoga

Exclusion Criteria:

* non-students
* inappropriate for group therapy treatment
* physical injuries not appropriate for yoga participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-01; Primary Completion 2016-05 (Estimated); Study Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
Counseling Center Assessment of Psychological Symptoms-62 | change from baseline at 8 weeks
  Change in psychological symptoms from baseline on the Counseling Center Assessment of Psychological Symptoms-62 at 8 weeks is being assessed.
Outcome Questionnaire- 45.2 | change from baseline at 8 weeks
  Change in psychological symptoms from baseline on the Outcome Questionnaire- 45.2 at 8 weeks is being assessed.
Mindful Attention and Awareness Scale | change from baseline at 8 weeks
  Change in mindfulness from baseline on the Mindful Attention and Awareness Scale at 8 weeks is being assessed.